CLINICAL TRIAL: NCT05376371
Title: Health Systems Innovations for Supporting Transitions of Care for Incarcerated People Living With HIV, Hepatitis C, and Substance Use Disorder
Brief Title: Criminal Justice Coordinated Transitional Care
Acronym: CJC-TraC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0398; 1R01DA047889-01A1 (NIH); Protocol Version 6/9/2024 (Other: UW Madison); A534265 (Other: UW Madison)
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: HIV; Hepatitis C; Substance Use Disorders
Keywords: incarcerated; transition; release
MeSH Terms: conditions — Hepatitis C; Substance-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CJC-TraC Intervention (Experimental): Incarcerated individuals with HIV, hepatitis C, or substance use disorder readying for release will enroll in the CJC-TraC intervention intended to assist in transitioning their health care.
  Interventions: Other: CJC-TraC

INTERVENTIONS:
Other: CJC-TraC — CJC-TraC utilizes a nurse case manager (NCM) to coordinate the participant's transitional care through release from a correctional facility. The NCM will visit either in person or via telehealth with the participant up to 4 times while incarcerated, and up to 4 times after release.

SUMMARY:
This project aims to enroll 220 incarcerated individuals living with HIV, Hepatitis C (HCV), or history of substance misuse preparing for release into a pilot implementation study to test the feasibility and acceptability of an adapted Coordinated Transitional Care intervention in a Criminal Justice setting (CJC-TraC). Participants can expect to be on study for up to 6 months.

DETAILED DESCRIPTION:
This protocol describes the second, implementation phase of a 5-year NIH-funded research project designed to evaluate post-incarceration health care utilization and outcomes for underserved people living with HIV, HCV and substance use disorder.

In the first study phase, conducted from 2020-21, the investigators analyzed Wisconsin Medicaid data to characterize the baseline level of outpatient care utilization for adults during their first 6 months after release from prison, and conducted formative research necessary to adapt an existing transitional care intervention, called C-TraC, to support individuals leaving prison.

The current project aims to enroll participants in a pilot implementation study to test the feasibility and acceptability of the adapted intervention in a criminal justice setting, which has been given the name "CJC-TraC."

Participants will be enrolled from one of two institutions:

* men from Oakhill Correctional Institute (OCI)
* women from the Wisconsin Women's Correctional System (WWCS)

Primary Objectives: To evaluate the feasibility and acceptability of CJC-TraC when implemented in a state prison system.

Secondary Objectives: To gather preliminary evidence describing the effectiveness of CJC-TraC for improving the rate of outpatient care utilization.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and speak in English
* Plans to reside in Wisconsin after release
* Eligible for Wisconsin Medicaid and willing to enroll prior to release
* Has a history of one or more of the following: current HIV infection, current or past HCV infection, identified need for substance use related services based on Correctional Offender Management Profiling for Alternative Sanctions (COMPAS) assessment
* Anticipated release date (must be within 6 months of review)

Exclusion Criteria:

* Unable to provide informed consent form or impaired ability to make decisions
* Planned discharge to another correctional facility or other carceral setting (e.g. release to jail or immigration detention center)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Westergaard, MD, PhD, MPH, Principal Investigator — UW School of Medicine and Public Health
Locations (2):
- United States (2):
  - Oakhill Correctional Institution, Oregon, Wisconsin
  - Robert E. Ellsworth Correctional Center, Union Grove, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CJC-TraC Intervention
Started | 219
Completed | 209
Not Completed | 10
Not completed — change in release date | 10

BASELINE CHARACTERISTICS:
Arm/Group | CJC-TraC Intervention
Number analyzed (Participants) | 219
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 213
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: Years] | 41 [21 to 75]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 105
  Male | 112
  Unknown: Missing Data | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 203
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 57
  White | 121
  More than one race | 15
  Unknown or Not Reported | 13
Region of Enrollment [Number; unit: participants]
  United States | 219

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Outcome: Number of Participants Who Are Enrolled and Complete the Baseline Study Assessment
Description: The number who successfully enrolled and completed the baseline assessment demonstrates the feasibility of engaging the target population in the prison setting.
Time Frame: at enrollment, up to 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | CJC-TraC Intervention
Number analyzed (Participants) | 219
Participants | 219

2. Primary Outcome: Feasibility Outcome: Number of Pre-release CJC-TraC Intervention Sessions Completed With the Nurse Case Manager for Each Participant
Description: The investigators plan for 3 pre-release sessions with additional sessions as needed. The results will be reported in total and for each institution.
Time Frame: pre-release, up to 3 months
Population: All enrolled participants were eligible to receive pre-release intervention sessions
Measure: Mean (Standard Deviation); unit: sessions
Units Other Than Participants: pre-release sessions
Arm/Group | CJC-TraC Intervention
Number analyzed (Participants) | 219
Number analyzed (pre-release sessions) | 679
sessions | 3.1 (1.2)

3. Primary Outcome: Feasibility Outcome: Number of Post-release Telephone Contact Attempts Between the CJC-TraC Nurse Case Manager and Study Participants
Description: The investigators plan for 2 post-release sessions with additional sessions as needed.
Time Frame: post-release, up to 6 months
Population: Of 219 individuals enrolled in the study, 10 were withdrawn because of a change in their release date after enrollment. The 209 who were released from prison during the study period were evaluated for the study outcomes.
Measure: Mean (Standard Deviation); unit: telephone contact attempts
Units Other Than Participants: telephone contact attempts
Arm/Group | CJC-TraC Intervention
Number analyzed (Participants) | 209
Number analyzed (telephone contact attempts) | 1212
telephone contact attempts | 5.8 (3.7)

4. Primary Outcome: Feasibility Outcome: Number of Study Participants Who Are Retained in Follow-up for Three Months and Complete the End-of-study Assessment
Time Frame: within 3-months following release (up to 6 months on study)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CJC-TraC Intervention
Number analyzed (Participants) | 209
Participants | 158

5. Primary Outcome: Acceptability Measured by the Number of Study Participants Who Rated the Volume of Pre-release Intervention Sessions as Appropriate
Description: Of participants who enroll and complete a follow up assessment, percentage of participants who responded to questions soliciting their perspectives about the intervention usefulness.
Time Frame: within 3-months following release (up to 6 months on study)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CJC-TraC Intervention
Number analyzed (Participants) | 209
Participants | 116

6. Primary Outcome: Acceptability Measured by the Number of Study Participants Who Rated the Volume of Post-release Intervention Contacts as Appropriate
Description: as for outcome 5
Time Frame: within 3-months following release (up to 6 months on study)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CJC-TraC Intervention
Number analyzed (Participants) | 209
Participants | 123

7. Primary Outcome: Acceptability Measured by the Number of Department of Corrections (DOC) Staff Who Rated the Intervention Acceptable, Useful, or Appropriate
Time Frame: up to 3 months
Population: 5 Staff from the prison system responded to the feedback survey
Measure: Number; unit: staff members from prison system
Groups:
- CJC-TraC Intervention - WIDOC Staff Survey: A sample of employees of the prison where the intervention was pilot tested, comprised of those who voluntarily completed a short online survey to rate the favorability of the intervention.
Arm/Group | CJC-TraC Intervention - WIDOC Staff Survey
Number analyzed (Participants) | 5
staff members from prison system | 5

8. Primary Outcome: Acceptability Assessed by Subjective Experience of the Participant (Qualitative Measure) Reported Here as Number of Participants Completing Acceptability Interviews
Description: Exploratory results of qualitative interviews among a subset of intervention participants.
Time Frame: within 3-months following release (up to 6 months on study)
Population: In total, 30 individuals (15 men and 15 women) participated in interviews between April 2023 and December 2024
Measure: Count of Participants; unit: Participants
Arm/Group | CJC-TraC Intervention
Number analyzed (Participants) | 30
Participants | 30

9. Secondary Outcome: Attendance at Non-emergency Outpatient Care Visits Within 3-months Following Release
Description: Based on review of medical records and Wisconsin Medicaid claims data, the occurrence of outpatient medical care visits, not including emergency department or urgent care visits.
Time Frame: within 3-months following release (up to 6 months on study)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CJC-TraC Intervention
Number analyzed (Participants) | 209
Participants | 149

10. Secondary Outcome: Number Days Until the First Non-emergency Outpatient Visit Following Release, Reported Here as Number of Participants With Visits Occurring Within 60 Days
Time Frame: within 3-months following release (up to 6 months on study)
Measure: Count of Participants; unit: Participants
Arm/Group | CJC-TraC Intervention
Number analyzed (Participants) | 209
Participants | 141

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse event was defined as unexpected death from any cause that was reported to the study team during the 12 week follow-up period. Acute hospitalizations and emergency department visits were not considered adverse events because they are common in this population and represented one of the study outcomes.
Arm/Group | CJC-TRAC Intervention
All-Cause Mortality (participants affected / at risk) | 2/209
Serious Adverse Events (participants affected / at risk) | 0/209
Other Adverse Events (participants affected / at risk) | 0/209

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT05376371/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT05376371/ICF_000.pdf